CLINICAL TRIAL: NCT02335216
Title: A Post Market ObServational StudY on the Effect of DRG StiMulation in PATients witH Chronic Pain Following Surgical Lumbar DiscectomY (Failed Back Surgery Syndrome): SYMPATHY
Brief Title: A Post Market Study on Dorsal Root Ganglion (DRG) Stimulation in Failed Back Surgery Syndrome (FBSS)
Acronym: SYMPATHY
Status: Terminated | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-SMI-2013
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated Subjects: All subjects recruited and treated with the Axium neurostimulator
  Interventions: Device: Implantation with the commercially available Axium neurostimulator

INTERVENTIONS:
Device: Implantation with the commercially available Axium neurostimulator

SUMMARY:
18-SMI-2013 is a post market, observational, questionnaire based study to assess the effectiveness of the commercially available Axium neurostimulator in the management of chronic pain following lumbar discectomy (Failed Back Surgery Syndrome)

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Chronic pain following surgical lumbar discectomy for at least 6 months
4. Failed conservative treatments for chronic pain including but not limited to pharmacological therapy, physical therapy and interventional pain procedures for chronic pain
5. Minimum baseline pain rating of 60 mm on the Visual Analog Scale in the subjects primary area of pain
6. Subject is able to provide written informed consent

Exclusion Criteria:

1. Female subject of childbearing potential is pregnant/nursing or plans to become pregnant during the course of the study
2. Escalating or changing pain condition within the past month as evidenced by investigator examination
3. Subject has had corticosteroid therapy at an intended site of stimulation within the past 30 days
4. Subject has had radiofrequency treatment of an intended target Dorsal Root Ganglion within the past 3 months
5. Subject currently has an active implantable device including implantable cardioverter defibrillator, pacemaker, spinal cord stimulator or intrathecal drug pump
6. Subject is unable to operate the device
7. Subjects with indwelling devices that may pose an increased risk of infection
8. Subjects currently has an active infection
9. Subject has participated in another clinical investigation within 30 days
10. Subject has a coagulation disorder or uses anticoagulants that, in the opinion of the investigator, precludes participation
11. Subject has been diagnosed with cancer in the past 2 years.
12. Subject has an anatomical spinal abnormality which is anticipated to require further surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from chronic pain post discectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St Antonius Ziekenhuis, Nieuwegein, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Subjects: All subjects enrolled into the study with intent to treat with the Axium Neurostimulator
Period: Overall Study
Arm/Group | All Enrolled Subjects
Started | 22
Received Trial System | 16
Received Permanent System | 13
Completed | 9
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 22
Age, Continuous [Mean (Full Range); unit: years] | 51 [26 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity for Overall Pain From Pre-treatment Baseline
Description: The Visual Analog Scale (VAS) is self-administered instrument assessing average pain intensity. Subjects rated their pain on a horizontal line, 10 cm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher pain level. The values range from 0 (minimum pain) to 10 (maximum pain).
Time Frame: Baseline, 3, 6 and 12 Months
Population: Differences in participants over time is due to early withdrawals and missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Subjected Treated With the Permanent Implantable Axium System: All subjects treated with the Axium implantable neurostimulator
Arm/Group | Subjected Treated With the Permanent Implantable Axium System
Number analyzed (Participants) | 13
units on a scale
  Baseline | 7.7 (1.1)
  3-Month Visit: number analyzed (Participants) | 9
  3-Month Visit | 2.9 (3.0)
  6-Month Visit: number analyzed (Participants) | 11
  6-Month Visit | 2.6 (3.6)
  12-Month Visit: number analyzed (Participants) | 9
  12-Month Visit | 2.4 (2.9)

2. Primary Outcome: Percentage of Subjects With at Least 50% Pain Reduction
Description: Percent of subjects with at least a 50% reduction. The Visual Analog Scale (VAS) is self-administered instrument assessing average pain intensity. Subjects rated their pain on a horizontal line, 10 cm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher pain level. The values range from 0 (minimum) to 10 (maximum).
Time Frame: 3, 6 and 12-Month Visits
Population: Differences in participants over time is due to early withdrawals and missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Subjected Treated With the Permanent Implantable Axium System
Number analyzed (Participants) | 13
Participants
  3-Month Visit: number analyzed (Participants) | 10
  3-Month Visit | 9
  6-Month Visit: number analyzed (Participants) | 10
  6-Month Visit | 8
  12-Month Visit: number analyzed (Participants) | 9
  12-Month Visit | 7

ADVERSE EVENTS:
Time Frame: All adverse events reported spontaneously by the subject or observed by the investigator or his staff were recorded from the time of enrollment to study completion or early withdrawal.
Description: All-cause mortality was not assessed in this study.
Arm/Group | All Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 7/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=22)
Abdominal pain (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=22)
IPG Pocket Pain (Injury, poisoning and procedural complications) | 1 (1)
Buzzing noise in left ear (Ear and labyrinth disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Irritated ganglion (Nervous system disorders) | 1 (1)
Loss of stimulation (Injury, poisoning and procedural complications) | 1 (1)
Wound Infection (Infections and infestations) | 2 (2)
Dural puncture (Injury, poisoning and procedural complications) | 3 (3)
Hematoma/Infection (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days